CLINICAL TRIAL: NCT03245775
Title: A Randomized-controlled Trial to Compare the Reach, Effectiveness and Maintenance of Two Family-based Childhood Obesity Treatment Programs in a Medically Underserved Region
Brief Title: A Trial of Two Family-based Childhood Obesity Treatment Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of Nebraska (Other); Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jamie Zoellner, PhD RD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19748
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Childhood
Keywords: health disparities; community-based participatory research
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iChoose (Experimental): 12 bi-weekly sessions & 24 IVR calls/12 months, 24 physical activity sessions over 6 months; delivers intervention to parents and children only
  Interventions: Behavioral: iChoose
- Family Connections (Experimental): 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only
  Interventions: Behavioral: Family Connections

INTERVENTIONS:
Behavioral: iChoose — 12 bi-weekly sessions & 24 IVR calls/12 months, 24 physical activity sessions over 6 months; delivers intervention to parents and children only
  Arms: iChoose
Behavioral: Family Connections — 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only
  Arms: Family Connections

SUMMARY:
The primary aim is to determine the relative effectiveness in child BMI z-scores at 3, 6, and 12-months post baseline of iChoose+ versus Family Connections. Secondary aims are to determine (1) ongoing reach, fidelity, and implementation costs, (2) community capacity for implementation and sustainability, (3) relative impact on family eating/physical activity and parental weight, and (4) relative adherence and potential dose response relationships.

DETAILED DESCRIPTION:
In partnership with the Community Advisory Board and Parent Advisory Team, with a goal to improve the magnitude of weight reductions and increase the likelihood of iChoose sustainability in the community, the investigators propose to test iChoose+ that will (1) extend iChoose to a 6-month program, followed by 12 bi-weekly maintenance telephone calls, congruent with the 12-month Bright Bodies program duration, (2) formalize a Parent Health Advisory model of previous iChoose families to serve as a 'peer support safety net' for new program participants, and (3) deliver support calls using interactive voice response (IVR) automation to reduce the burden on community stakeholder implementation. When reflecting on and interpreting the outcomes of the previous planning grant, the Community Advisory Board and Parent Advisory Team also identified the need to use a study design that allowed all participants the opportunity to benefit and, with this in mind, to test alternative family-based childhood obesity program options that improve reach within the broad Dan River Region population of minority, low-income, and geographically dispersed families. Thus, the Community Advisory Board and Parent Advisory Team returned to a potential option for delivery that was considered earlier in the planning grant process and was rated highly for scalability- Family Connections, an adaptation of Golan's Home Environmental Change model that focuses exclusively on parents as the agents of change. When compared to iChoose+ (12 bi-weekly sessions & 24 IVR calls/12 months), Family Connections has fewer sessions and fewer IVR support calls over a shorter period of time (2 in-person sessions spaced one week apart & 10 IVR calls/6 months), delivers intervention to parents only, and promotes physical activity, but does not include structured exercise sessions. Still, in previous studies Family Connections led to significant reductions in child weight status, though smaller in magnitude than Bright Bodies, that were sustained 6-month post intervention completion. Committed to the goal of allowing all participating families an opportunity to benefit from study participation and the need for a sustainable family-based childhood obesity option, the Community Advisory Board and Parent Advisory Team propose a comparative effectiveness trial where eligible families will be randomly assigned to: (1) iChoose+ (n=87) or to (2) Family Connections (n=87). Given the need to optimize program enrollment, participation, and retention in each program, both iChoose+ and Family Connections will include Parent Health Advisor support63-68 as refined by the Parent Advisory Team. The primary aim is to determine the relative changes in child BMI z-scores at 6 months post baseline of iChoose+ versus Family Connections, though additional assessments will occur at 3 and 12 months post baseline. Secondary aims include (1) determine ongoing reach, fidelity, and costs of implementation, (2) assess community capacity to implement and sustain childhood obesity programs, (3) determine impact on family eating and physical activity and parental weight by intervention, and (4) assess the adherence by intervention and potential dose response relationships. The primary study hypotheses are: (a) children in both conditions will reduce BMI-z scores significantly, when compared to baseline at 3, 6 and 12 months, but iChoose+ reductions will be significantly larger than Family Connections, (b) reach-the sample will be representative of the eligible regional population on demographic and behavioral factors, (c) implementation-the intervention components will be delivered with high fidelity in both conditions, but costs will be lower for Family Connections, (d) maintenance-a sustainability action plan will be completed to include strategies for continued delivery of iChoose+ and/or Family Connections (outcome dependent), (e) parent weight, parent/child behaviors, & tertiary outcomes that follow the same patterns as BMI z-scores, and (f), community capacity for implementing and sustaining a locally relevant FBCO treatment and maintenance program will remain high over time.

ELIGIBILITY:
Inclusion Criteria:

* Parent/child dyads will be eligible for participation if they reside in the Dan River Region

  * English speaking
  * child with a BMI percentile ranking of 85 or higher

    * Cohort 3 age eligibility changed from 8-12 to 5-15

Exclusion Criteria:

* children with a major cognitive impairment and parents or children with a medical contraindication for moderate physical activity.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zoellner JM, You W, Hill JL, Brock DP, Yuhas M, Alexander RC, Price B, Estabrooks PA. A comparative effectiveness trial of two family-based childhood obesity treatment programs in a medically underserved region: Rationale, design & methods. Contemp Clin Trials. 2019 Sep;84:105801. doi: 10.1016/j.cct.2019.06.015. Epub 2019 Jun 28. PMID 31260792

RESULTS

PARTICIPANT FLOW:
Groups:
- iChoose-Parent; iChoose-Child: 12 bi-weekly sessions & 24 IVR calls/12 months, 24 physical activity sessions over 6 months; delivers intervention to parents and children only
  iChoose: 12 bi-weekly sessions & 24 IVR calls/12 months, 24 physical activity sessions over 6 months; delivers intervention to parents and children only
- Family Connections-Parent: 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only
  Family Connections: 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only
- Family Connections-Child: 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only. Children are enrolled and assessed at baseline and 6 months.
  Family Connections: 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only. Children are enrolled and assessed at baseline, 3 months, and 6 months.
Period: Overall Study
Arm/Group | iChoose-Parent | iChoose-Child | Family Connections-Parent | Family Connections-Child
Started | 66 | 70 | 62 | 69
Completed | 41 | 44 | 46 | 53
Not Completed | 25 | 26 | 16 | 16
Not completed — Lost to Follow-up | 25 | 26 | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Family Connections-Child: 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only
  Family Connections: 2 in-person sessions spaced one week apart & 10 IVR calls/6 months, promotes physical activity but does not include structured exercise sessions; delivers intervention to parents only
- Total: Total of all reporting groups
Arm/Group | iChoose-Parent | iChoose-Child | Family Connections-Parent | Family Connections-Child | Total
Number analyzed (Participants) | 66 | 70 | 62 | 69 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 70 | 0 | 69 | 139
  Between 18 and 65 years | 66 | 0 | 61 | 0 | 127
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (7.2) | 10.1 (1.7) | 39 (9.6) | 10.0 (1.7) | 10.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 46 | 60 | 34 | 204
  Male | 2 | 24 | 2 | 35 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 13 | 3 | 6 | 25
  Not Hispanic or Latino | 63 | 57 | 59 | 63 | 242
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 33 | 31 | 29 | 31 | 124
  White | 32 | 35 | 30 | 31 | 128
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 3 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 66 | 70 | 62 | 69 | 267
BMI status [Count of Participants; unit: Participants] — For children Body Mass Index (BMI) is a percentile generated from gender and age specific height and weight charts. A BMI percentile less than 85% is normal, 85-94% is overweight, and 95% or greater is considered obese.
  For adults, BMI is determined through height and weight ratios. Normal BMI is 18.5-24.9; Overweight is 25-29.9, and Obese is 30 or greater.
  Participants
    Normal | 8 | 0 | 1 | 0 | 9
    Overweight | 9 | 20 | 12 | 21 | 62
    Obese | 49 | 50 | 49 | 48 | 196
Health Insurance Type [Count of Participants; unit: Participants]
  Medicaid | 19 | 41 | 20 | 45 | 125
  Private | 35 | 25 | 28 | 21 | 109
  None | 6 | 2 | 6 | 1 | 15
  Medicare | 2 | 0 | 5 | 0 | 7
  Other | 4 | 2 | 3 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Child Body Mass Index (BMI) Z-score at 6 Months
Description: child BMI is converted to a BMI Z score which uses a standardized distribution. A BMI z score of 0 indicates an average BMI for the childs height, weight, age, and gender. Positive z-scores indicate the number of standard deviations above the norm, while negative numbers indicate the number of standard deviations below the norm. Higher z scores indicate a greater BMI status for the child. The primary outcome is a change score, or the difference between the 6 month BMI z-score and the Baseline BMI z-score. A negative score will indicate BMI z score status reductions and is a positive finding.
Time Frame: Baseline and 6-months
Measure: Mean (95% Confidence Interval); unit: z-scores
Arm/Group | iChoose-Child | Family Connections-Child
Number analyzed (Participants) | 70 | 69
z-scores | 0.03 [-0.13 to 0.19] | 0.00 [-0.16 to 0.16]

2. Secondary Outcome: Change From Baseline of Parent Body Mass Index (BMI) at 6 Months
Description: BMI is the persons weight divided by the square of their height. BMI categories help to classify individuals as underweight (less than 18.5), normal (18.5-24.9), overweight (25-29.9), and obese (30 or higher). Parent BMI change scores are the difference between the 6 month calculated BMI and the Baseline BMI. Negative scores indicate improvement in BMI status over this 6 month period.
Time Frame: Baseline and 6-months
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | iChoose-Parent | Family Connections-Parent
Number analyzed (Participants) | 66 | 62
kg/m^2 | -1.04 [-4.15 to 2.08] | 0.04 [-2.95 to 3.02]

3. Secondary Outcome: Change From Baseline in the Pediatric Quality of Life Inventory for Children Score at 6 Months
Description: The Pediatric Quality of Life Inventory is a 23-item instruments that assesses four domains of health (physical, emotional, social, and school functioning). Scoring is reported as a percent (0-100), higher scores indicate better health related quality of life. The change score is calculated as the difference between the 6 month and baseline scores. A positive difference is considered an improvement in quality of life.
Time Frame: Baseline and 6-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iChoose-Child | Family Connections-Child
Number analyzed (Participants) | 70 | 69
score on a scale | -0.7 [-7.3 to 5.9] | 5.0 [-0.5 to 10.4]

4. Secondary Outcome: Change From Baseline in the Healthy Days Core Module for Parents at 6 Months
Description: The Healthy Days Core Module is a measure of quality of life through self reports of the total number of physical and mental health "sick days" (e.g., unable to do daily activities) in the past month. Higher scores indicate more unhealthy days, or lower quality of life. Change scores are calculated as the difference between 6 month and baseline scores. A negative change score indicates a decrease in unhealthy days and thereby and increase in quality of life.
Time Frame: Baseline and 6-months
Measure: Mean (95% Confidence Interval); unit: number of unhealthy days in past month
Arm/Group | iChoose-Parent | Family Connections-Parent
Number analyzed (Participants) | 66 | 62
number of unhealthy days in past month | 3.1 [-1.4 to 7.5] | -3.8 [-8.2 to 0.5]

ADVERSE EVENTS:
Time Frame: From baseline enrollment, through the 12-month f/u period.
Arm/Group | iChoose-Parent | iChoose-Child | Family Connections-Child | Family Connections-Parent
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/70 | 0/69 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/70 | 0/69 | 0/62
Other Adverse Events (participants affected / at risk) | 0/66 | 0/70 | 0/69 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT03245775/Prot_SAP_000.pdf